CLINICAL TRIAL: NCT07203430
Title: Assessing Adaptations in Biopsychosocial Factors and Muscle Morphology After a Resistance Exercise Intervention in Individuals With Low Back Pain
Brief Title: Biopsychosocial Factors and Muscle Morphology After a Resistance Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Abigail Wilson, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12
Record Dates: First submitted 2025-09-22; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain, Chronic
Keywords: Exercise; Low Back Pain
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): During visits 2-13, participants will attend 2-3 sessions per week, with a minimum of 48 hours between visits, and must complete all study visits 6 weeks after enrollment. Participants in the intervention group will perform 3 sets of low back extension exercise on the Roman chair until volitional exhaustion. The three sets will be performed to volitional exhaustion or 20 repetitions, whichever comes first. If more than 20 repetitions can be completed after a set the investigator will add resistance according to the NSCA's guidelines (2.5-10% increase).
  Interventions: Other: 45-Degree Roman Chair Exercise
- Control Group (No Intervention): Participants in the control group will not complete the low back extension exercise and will be told to continue activity as usual. All participants will complete a training log and detail the type of resistance exercise performed, the number of sets and repetitions completed, and the weight used.

INTERVENTIONS:
Other: 45-Degree Roman Chair Exercise — Participants in the intervention group will perform 3 sets of low back extension exercise on the Roman chair until volitional exhaustion. The three sets will be performed to volitional exhaustion or 20 repetitions, whichever comes first. If more than 20 repetitions can be completed after a set the investigator will add resistance according to the NSCA's guidelines (2.5-10% increase).
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to evaluate the longitudinal effects of a four-week dynamic resistance training program using the 45-degree Roman chair on pain sensitivity changes after exercise and lumbar muscle performance in individuals with chronic low back pain (LBP). This study will consist of three specific aims. Aim 1 examines changes in local exercise-induced hypoalgesia. Aim 2 will assess changes in lumbar multifidus and erector spinae thickness using ultrasound imaging before and after the intervention. Aim 3 will evaluate changes in lumbar extensor strength (handheld dynamometry (HHD)) and endurance (Biering-Sørensen test).

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain lasting ≥ 12 weeks
* current pain intensity ≥ 3/10 but no higher than an 8/10 on the Numeric Pain Rating Scale (NPRS) within the past 48 hours
* resistance trained (defined as 2x/week for the past 8-12 weeks)
* able to read and speak English for informed consent and completion of questionnaires
* willing and physically able to complete all testing and intervention sessions.

Exclusion Criteria:

* History of spinal surgery, fusion, or fracture within the past 6 months
* diagnosed degenerative disc disease, scoliosis, or spinal pathology that precludes safe exercise participation
* use of an assistive device for walking (cane, walker) within the past year
* pregnancy, due to contraindications for exercise testing and ultrasound -body weight ≥ 300 lbs., which exceeds the safe capacity of the Roman chair --
* current tobacco/nicotine use
* current enrollment in physical therapy or structured rehabilitation for LBP,
* cardiovascular, pulmonary, metabolic, or systemic disease that increases risk during exercise
* nociplastic pain conditions (e.g., fibromyalgia) or neurological conditions that confound EIH responses
* inability to complete ≥ 8 Roman chair repetitions with proper form during screening
* non-English speaking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Exercise Induced Hypoalgesia | Weeks 1 and 4
  Participants will perform one set of back extension exercise on a 45-degree Roman chair until volitional exhaustion. Pressure Pain Threshold applied over the low back will be examined before and after exercise.
Muscle Thickness | Weeks 1 and 4
  Ultrasound imaging to assess muscle thickness of the erector spinae and the multifidus muscles will be completed.
Muscle Strength | Weeks 1 and 4
  Back extensor strength will be assessed using maximal voluntary isometric contraction of the back extensor muscles using a handheld dynamometer.
Muscle Endurance | Weeks 1 and 4
  The Biering-Sorensen test will be performed in which participants lie prone on a treatment table with the lower body secured to the table. Participants will be instructed to cross their arms over their chest and maintain their torso in a horizontal position with the upper body unsupported, parallel to the floor.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No